CLINICAL TRIAL: NCT03880513
Title: Cardiovascular Status in Patients With Endogenous Cortisol Excess (Cushing's Syndrome)
Acronym: CV-CORT-EX
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CV-CORT-EX
Record Dates: First submitted 2018-07-12; First posted 2019-03-19 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Endogenous Cushing's Syndrome
Keywords: Endogenous Cushing's Syndrome; Cardiovascular status; Metabolic profile; Endothelial function; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Longitudinal study: Patients during overt and after cure of endogenous Cushing's syndrome.
  Interventions: Diagnostic Test: Cardiovascular status and quality of life
- Cross-sectional study: Patients with proven endogenous Cushing's syndrome (overt or subclinical).
  Interventions: Diagnostic Test: Cardiovascular status and quality of life

INTERVENTIONS:
Diagnostic Test: Cardiovascular status and quality of life — Psychosocial and cardiovascular evaluation includes medical history, physical examination, laboratory tests, analysis of endothelial function, 24h blood pressure profile, Holter ECG, transthoracic echocardiography, cardiac MRI, and quality of life assessment

SUMMARY:
Within this trial, the cardiovascular and mental status as well as the metabolic profiles of patients with endogenous cortisol excess are evaluated.

DETAILED DESCRIPTION:
Endogenous Cushing's syndrome (CS) is associated with increased cardiovascular (CV) morbidity and reduced general health status. It has been shown that these impairments may be reversible after cure of hypercortisolism. However, previous studies were restricted to selected CV aspects.

The primary aim of the CV-CORT-EX study is to comprehensively assess left ventricular function and morphology of patients with endogenous CS. Secondly, we examine long-term changes of CV function, endothelial function, psychosocial status, bio-impedance, and quality of life.

Within the longitudinal study, patients will be investigated at initial diagnosis and at least 6 months after cure of CS. Within the cross-sectional study, we aim to comprehensively phenotype patients with endogenous CS and unknown CV disease. Results will finally be compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Cross-sectional study:History of clinically and biochemically proven endogenous Cushing's syndrome (overt or subclinical)
* Longitudinal study: Patients with clinically and biochemically proven endogenous Cushing's syndrome (initial diagnosis or recurrent disease)

Exclusion Criteria:

* Glucocorticoid pharmacotherapy for >12 months within the previous 3 years
* Structural heart disease, chronic heart failure (>NYHAII), systemic or single organ disease potentially affecting cardiac function
* Arterial hypertension (uncontrolled with >3 antihypertensive drugs)
* Pregnancy
* Drug abuse
* Cardiac Magnetic Resonance Imaging (cMRI) substudy: patients with renal failure are excluded from the cMRI study (MDRD <60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross-sectional study:
  - History of clinically and biochemically proven endogenous Cushing's syndrome (overt or subclinical)
  Longitudinal study:
  - Patients with clinically and biochemically proven endogenous Cushing's syndrome (initial diagnosis or recurrent disease)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular status - pathological cardiac MRI | 7 years
  Number of patients with pathological results (ejection fraction (<55%), pericardial effusion, thrombus, adipose tissue, perfusion defects, late enhancement, valvular or wall motion abnormalities).

SECONDARY OUTCOMES:
Cardiovascular status - pathological cardiac echocardiography | 7 years
  Characterization of left ventricular (LV) morphology and function, assessment of diastolic function and systolic strain. Assessment of regional and global LV function, characterization of right ventricular systolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, Professor, Study Director — University Hospital Wuerzburg
Locations (1):
- University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kamenicky P, Redheuil A, Roux C, Salenave S, Kachenoura N, Raissouni Z, Macron L, Guignat L, Jublanc C, Azarine A, Brailly S, Young J, Mousseaux E, Chanson P. Cardiac structure and function in Cushing's syndrome: a cardiac magnetic resonance imaging study. J Clin Endocrinol Metab. 2014 Nov;99(11):E2144-53. doi: 10.1210/jc.2014-1783. Epub 2014 Aug 5. PMID 25093618
- [Derived] Ehrlich K, Morbach C, Reiter T, Heuschmann PU, Hannemann A, Fassnacht M, Stork S, Hahner S, Deutschbein T. Rationale and design of the cardiovascular status in patients with endogenous cortisol excess study (CV-CORT-EX): a prospective non-interventional follow-up study. BMC Endocr Disord. 2021 Jan 8;21(1):11. doi: 10.1186/s12902-020-00665-7. PMID 33419423